CLINICAL TRIAL: NCT04115553
Title: Assessment of Venous Drainage in Idiopathic Intracranial Hypertension
Acronym: HYPERPIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2019_843_0056
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Hypertension
Keywords: Intracranial Hypertension; venous drainage; MRI; blood flow; cerebrospinal fluid flow
MeSH Terms: conditions — Intracranial Hypertension | interventions — Magnetic Resonance Imaging; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- idiopathic intracranial hypertension (Experimental): patients with idiopathic intracranial hypertension
  Interventions: Diagnostic Test: MRI examination; Diagnostic Test: ECG
- healthy subjects (Sham Comparator): Healthy subjects
  Interventions: Diagnostic Test: MRI examination; Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: MRI examination — Subjects will be placed in supine position. The systematic use of a headset will reduce the noise inherent to the machine. Standard MRI examination using a 32-channel head coil consists of angiographic, morphological and phase-contrast 2D flow sequences. The flow planes are set perpendicularly to the structure axis (blood or CSF regions). The velocity measured in the pixels inside the region of interest allow the calculation of a mean flow rate as well as the volume displaced during a cardiac cycle.
  Other Names: Magnetic resonance imaging (MRI)
Diagnostic Test: ECG — A cardiac synchronization system using peripheral ECG allows the synchronization with the subject's heart rate.
  Other Names: Electrocardiogram

SUMMARY:
Intracranial hypertension (IIH) is a disorder producing a syndrome of increased intracranial pressure secondary to a compressive intracranial lesion or said to be idiopathic. The most common symptoms are headaches, blindness, pulsatile tinnitus or papillary edema. There are many options for the treatment of IIH, especially neurosurgery (derivation of cerebrospinal fluid or stent placement). Currently, idiopathic IIH has no clear etiology but the hypothesis of sino-venous insufficiency is more and more recognized. The assumption of venous insufficiency has not been demonstrated so far. Therefore the investigators propose to demonstrate that cerebral venous drainage pathways are altered in adult patients with idiopathic intracranial hypertension in comparison to healthy individuals having normal circulation. Assessment will be performed using Magnetic Resonance Imaging which is part of the patient care.

DETAILED DESCRIPTION:
The investigator working hypothesis is an impairment of the cerebral venous drainage in IIH compared to the circulation observed in healthy volunteers considered as the reference. The research will focus on adult patients referred to the imaging department for intracranial hypertension assessment. MRI support is common for this type of request The reference will be established in a population of healthy volunteers for whom MRI blood flow measurements will be performed. In addition to the primary objective, the investigators assess the impact of IIH on CSF dynamics The study does not present any risk for the subject, any contraindication to MRI examination being respected. The subjects will undergo MRI examination including morphological and flow sequences without contrast injection. The flow sequences, in planes located at the C2-C3 and aqueductal levels, will be used to measure vascular flows (venous and arterial) and CSF oscillatory volumes. Image post-processing will be performed on a semi-automatic software allowing to extract fluid dynamics parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age : >18 years old
* adult patients referred to the imaging department for intracranial hypertension assessment
* adult control subjects without history of cerebral or vascular pathology

Exclusion Criteria:

* history of cerebral or vascular pathology for the control subjects
* pregnant woman
* claustrophobia
* major obesity
* any contraindication to MRI exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Ratio between jugular vein flow and total arterial brain flow. | day 0 = day of inclusion
  Venous jugular flow is the sum right and left internal jugular vein flows. Total arterial flow is the sum of right and left internal carotid and vertebral arteries flows.

SECONDARY OUTCOMES:
CSF (cerebrospinal fluid) Stroke volumes | day 0 = day of inclusion
  CSF oscillatory volumes measured at the Sylvius' aqueduct and sub-arachnoidian space levels

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No